CLINICAL TRIAL: NCT06239714
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, SAD and MAD Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneously Administered SGB-3403 in Healthy Volunteers and Subjects With Elevated LDL-C
Brief Title: A Study to Evaluate SGB-3403 in Healthy Volunteers and Subjects With Elevated Low-Density Lipoprotein Cholesterol (LDL-C)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Suzhou Sanegene Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGB-3403-001
Record Dates: First submitted 2024-01-08; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Hyperlipidemias
MeSH Terms: conditions — Hyperlipidemias | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- SGB-3403(SAD) (Experimental)
  Interventions: Drug: SGB-3403
- placebo(SAD) (Placebo Comparator)
  Interventions: Other: Placebo
- SGB-3403(Non-Statin MAD) (Experimental)
  Interventions: Drug: SGB-3403
- placebo(Non-Statin MAD) (Placebo Comparator)
  Interventions: Other: Placebo
- SGB-3403 and atorvastatin(statin MAD) (Experimental)
  Interventions: Drug: SGB-3403; Other: Atorvastatin
- placebo and atorvastatin(statin MAD) (Placebo Comparator)
  Interventions: Other: Atorvastatin; Other: Placebo

INTERVENTIONS:
Drug: SGB-3403 — SGB-3403 is a synthetic, chemically modified small interfering ribonucleic acid (siRNA) targeting proprotein convertase subtilisin kexin type 9 (PCSK9) messenger ribonucleic acid (mRNA) with a covalently attached triantennary N-acetylgalactosamine (GalNAc) ligand.
  Arms: SGB-3403 and atorvastatin(statin MAD); SGB-3403(Non-Statin MAD); SGB-3403(SAD)
Other: Atorvastatin — The dosage of atorvastatin was determined by the investigator
  Arms: SGB-3403 and atorvastatin(statin MAD); placebo and atorvastatin(statin MAD)
Other: Placebo — Normal saline 0.9%
  Arms: placebo and atorvastatin(statin MAD); placebo(Non-Statin MAD); placebo(SAD)

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, single ascending dose (SAD) and multiple ascending doses (MAD) of SGB-3403 when single administered subcutaneously to healthy volunteers and multiple administered subcutaneously to subjects with elevated LDL-C to evaluate the safety, tolerance, PK, and PD.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, single ascending dose (SAD) and multiple ascending doses (MAD) of SGB-3403 when single administered subcutaneously to healthy volunteers and multiple administered subcutaneously to subjects with elevated LDL-C. The study will be performed in 2 phases: SAD and MAD.

ELIGIBILITY:
Inclusion Criteria in SAD:

* Male and female subjects aged 18 to 55 years are included.
* Body mass index between 19 and 32 kg/m2, inclusive.
* Physical examination, vital signs, 12-lead electrocardiogram, and laboratory tests will be normal or slightly abnormal but not clinically significant according to the Investigator's judgment.
* Willing to comply with the protocol required visit schedule and visit requirements and provide written informed consent.

Exclusion Criteria in SAD:

* An underlying known disease or surgical or medical condition that, in the opinion of the Investigator, might interfere with the interpretation of the clinical study results.
* The positive result of hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), human immunodeficiency virus (HIV) antibody, or syphilis at screening.
* Alanine aminotransferase (ALT), total bilirubin (TBIL), aspartate aminotransferase (AST), alkaline phosphatase (ALP), or gamma-glutamyl transferase (GGT) > 1.5 × ULN (upper limit of normal).
* Serum creatinine exceeds the upper limit of normal at screening.
* History of multiple drug allergies or allergic reactions to an oligonucleotide or N acetylgalactosamine (GalNAc).
* History of intolerance to subcutaneous (SC) injection or relevant abdominal scarring (surgical, burns, etc.)
* Received an investigational agent within 28 days or 5 half-lives (whichever is longer) before the first dose of the study drug or are in another clinical study, received INCLISIRAN within 1 year.
* Use any Chinese herbs, vitamins, or supplements known to affect lipid metabolism (e.g., fish oil > 1000 mg/ day, medicines, or health products containing red yeast rice) within 28 days before receiving the test drug.
* Any conditions which, in the opinion of the Investigator, would make the subject unsuitable for enrollment or could interfere with the subject's participation in or completion of the study.

Inclusion Criteria in MAD:

* Male and female subjects aged 18 to 65 years are included.
* Body mass index between 19 and 35 kg/m2, inclusive.
* Serum LDL-C ≥ 2.6mmol/L (≤ 100 mg/dL) and ≤ 4.9 mmol/L (≤ 190 mg/dL) at screening.
* Fasting triglyceride < 4.52 mmol/L (< 400 mg/dL) at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-02-18 (Estimated); Primary Completion 2025-02-18 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | 57 days
  To evaluate the safety and tolerability of SGB-3403 when administered subcutaneously as a single dose to healthy volunteers
Number of participants with abnormal laboratory tests results | 57 days
  To evaluate the safety and tolerability of SGB-3403 when administered subcutaneously as a single dose to healthy volunteers
Number of participants with adverse events (AEs) | 169 days
  To evaluate the safety and tolerability of SGB-3403 when administered subcutaneously in multiple-dose to subjects with elevated LDL-C
Number of participants with abnormal laboratory tests results | 169 days
  To evaluate the safety and tolerability of SGB-3403 when administered subcutaneously in multiple-dose to subjects with elevated LDL-C

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | 48 hours
  To characterize the pharmacokinetics of SGB-3403 in healthy volunteers and subjects with elevated LDL-C
Area under the concentration-time curve (AUC) | 48 hours
  To characterize the pharmacokinetics of SGB-3403 in healthy volunteers and subjects with elevated LDL-C
LDL-C change from baseline | 180 days
  To evaluate the pharmacodynamic effect of SGB-3403 on serum levels of LDL-C in healthy volunteers
LDL-C change from baseline | 265 days
  To evaluate the pharmacodynamic effect of SGB-3403 on serum levels of LDL-C in subjects with elevated LDL-C
PCSK9 change from baseline | 180 days
  To evaluate the pharmacodynamic effect of SGB-3403 on plasma levels of proprotein convertase subtilisin/kexin type 9 in healthy volunteers
PCSK9 change from baseline | 265 days
  To evaluate the pharmacodynamic effect of SGB-3403 on plasma levels of proprotein convertase subtilisin/kexin type 9 in subjects with elevated LDL-C